CLINICAL TRIAL: NCT00129142
Title: A Randomized, Double Blind, Placebo Controlled, Multicenter Efficacy and Safety Study of Toremifene Citrate for Prevention of Bone Fractures in Men With Prostate Cancer on Androgen Deprivation Therapy
Brief Title: Toremifene Citrate for Prevention of Bone Fractures in Men With Prostate Cancer on Androgen Deprivation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GTx (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: G300203
Record Dates: First submitted 2005-08-09; First posted 2005-08-11 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Prostate Cancer; Osteoporosis; Fractures
Keywords: Prostate cancer; Bone Loss; Osteoporosis; Fractures; Androgen Deprivation Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Osteoporosis; Fractures, Bone; Bone Diseases, Metabolic | interventions — Toremifene

INTERVENTIONS:
Drug: Toremifene Citrate

SUMMARY:
Androgen deprivation therapy (ADT) treatment for prostate cancer decreases the natural hormone called testosterone. This type of therapy is very effective for the treatment of prostate cancer. However, one of the side effects is bone loss or thinning of the bones that can lead to osteoporosis and an increased risk of bone fractures (breaking of the bones). The purpose of the study is to determine whether or not the addition of toremifene citrate (the study drug) to therapy can prevent or decrease the number of bone fractures and to evaluate its impact on side effects associated with testosterone reduction therapy.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in this study, subjects must meet all of the following criteria (minor deviations may be discussed with the medical monitor for possible inclusions):

* Give voluntary, signed informed consent in accordance with institutional policies
* Be male, aged ≥ 50 years
* Have histologically documented prostate cancer. Subjects with metastatic prostate cancer may still be considered for the study as long as they are not disqualified by other inclusion/exclusion criteria and there is a reasonable expectation that their medical condition will not interfere with the objectives of the study and that adequate follow-up and compliance with the study protocol can be achieved for the full 24-month duration of the study.
* Have been on:

  * ADT treatment (either luteinizing hormone-releasing agonist [LHRHa] or orchiectomy) for at least 6 months; Or
  * Intermittent LHRHa for at least the preceding 12 months is acceptable, but subjects must be maintained on uninterrupted treatment for the duration of this study once they are randomized into the study.
* Be aged ≥ 70 years or have BMD of lumbar spine or femoral neck at or below the specified thresholds for study entry:

  * Hologic BMD (g/cm2): L1-L4 - 0.926; Femoral neck - 0.717
  * Lunar BMD (g/cm2): L1-L4 - 1.050; Femoral neck - 0.840
* Serum prostate-specific antigen (PSA) ≤ 4 ng/mL
* Have a Zubrod performance status ≤ 1
* Subject weight < 300 lbs (weight limitation of DEXA equipment)
* Agree to complete a daily diary of medication intake and to provide tablet containers for accurate counts
* Agree to use an effective method of contraception, if the partner is of childbearing age, while on study
* Have adequate bone marrow, liver and renal function:

  * White blood cell (WBC) count ≥ 3,000/mm3;
  * Platelet count ≥ 100,000/mm3;
  * Bilirubin ≤ 1.5 mg/dL;
  * AST and ALT < 2x upper limit of normal;
  * Serum creatinine ≤ 2.0 mg%.

Exclusion Criteria:

Subjects with any of the following will not be eligible for enrollment:

* Taking bisphosphonates, selective estrogen receptor modulators (SERMs), parathyroid hormone (PTH), Forteo® (teriparatide), calcitonin, or oral glucocorticoids within 45 days of randomization
* Have any disease or condition that would preclude an accurate evaluation of radiographs of the thoracic and lumbar spine (at least eight evaluable vertebrae in the range T4 to L4) [for example, severe scoliosis, or sequelae of orthopedic procedures or other surgery]
* Have > 4 vertebral fragility fractures
* Have any history of other carcinomas within the last 5 years (except nonmelanoma cutaneous malignancies and superficial bladder cancer with no evidence of recurrence which will not be excluded). NOTE: Patients with cancers other than nonmelanoma cutaneous malignancies and superficial bladder cancer with no evidence of tumor recurrence for at least 5 years after definitive treatment will not be excluded from this study.
* Have Paget's disease of bone
* Have active systemic viral, bacterial or fungal infections requiring treatment
* Have, in the judgment of the investigator, a clinically significant concurrent illness or psychological, familial, sociological, geographical or other concomitant condition that would not permit adequate follow-up and compliance with the study protocol for the full 24-month duration of the study
* Received treatment with other investigational agents within 30 days prior to randomization
* Taking finasteride (e.g., Proscar®), dutasteride (e.g., Avodart®), Danocrine® (danazol) or testosterone-like supplements, such as dehydroepiandrosterone (DHEA) [subject is eligible if he stops these agents for a total washout of 45 days prior to randomization and agrees not to use these agents for the duration of the study]
* Taking herbal medicine or dietary supplements for prostate health, such as PC SPES and saw palmetto (also known as Serenoa repens) [subject is eligible if he stops these agents for a total washout of 45 days prior to randomization and agrees not to use these agents for the duration of the study]. Lycopene and selenium are not prohibited and no washout is required.
* Have a history of thromboembolic disease including deep vein thrombosis or pulmonary embolus
* Have a history of chronic hepatitis or cirrhosis
* Have received prior treatment with toremifene

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200
Dates: Start 2003-10; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects at 24 months with at least one new vertebral fracture determined by blinded central review of radiographs of the thoracic and lumbar spine

SECONDARY OUTCOMES:
Percentage of subjects with at least one new or worsening vertebral fracture at 24 months
Percentage of subjects with a clinical fragility fracture at 12 and 24 months
Percent change from baseline in lumbar bone mineral density (BMD) as measured by dual energy x-ray absorptiometry (DEXA) scan at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Steiner, M.D., Study Director — GTx
Locations (155):
- United States (136):
  - Urology Centers of Alabama, Homewood, Alabama
  - Coastal Clinical Research, Mobile, Alabama
  - Arkansas Urology, Little Rock, Arkansas
  - Advanced Urology Medical Center Clinical Trials, Anaheim, California
  - Urological Sciences Research Foudation, Culver City, California
  - Urological Associates of Central CA, Fresno, California
  - Center of Urologic Research, La Mesa, California
  - South Orange County Medical Research Center, Laguna Woods, California
  - Palo Alto VA, Palo Alto, California
  - San Bernadino Urological Associates, San Bernadino, California
  - Urological Physicians of San Diego, San Diego, California
  - Veterans Medical Research Foundation, San Diego, California
  - Pacific Clinical Research, Santa Monica, California
  - West Coast Clinical Research, Tarzana, California
  - Western Clinical Research, Inc., Torrance, California
  - Urology Associates, Denver, Colorado
  - Western Urological Research, Wheat Ridge, Colorado
  - Urologic Center, New Haven, Connecticut
  - Urological Associates of Bridgeport, Trumball, Connecticut
  - Connecticut Clinical Research, Waterbury, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - South Florida Medical Research, Aventura, Florida
  - Urology Consultants Inc., Clearwater, Florida
  - Atlantic Urological Associates, Daytona Beach, Florida
  - Urosearch, Inverness, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Advance Research Institute, New Port Richey, Florida
  - Central Florida Urology Group/ UroSearch, Ocala, Florida
  - Florida Foundation for Healthcare Research, Ocala, Florida
  - Winter Park Urology Associates, Orlando, Florida
  - Panama City Urology, Panama City Beach, Florida
  - Pinellas Urology, St. Petersburg, Florida
  - Southeastern Research Group, Tallahassee, Florida
  - Tampa Bay Urology, Tampa, Florida
  - UroSearch, Tavares, Florida
  - Cleveland Clinic-Florida, Weston, Florida
  - Midtown Urology, Atlanta, Georgia
  - Georgia Urology, Atlanta, Georgia
  - St. Joseph Research Institute, Atlanta, Georgia
  - Augusta VAMC, Augusta, Georgia
  - Southeastern Medical Research Institute, Columbus, Georgia
  - Urology Enterprises, Marietta, Georgia
  - Harbin Clinic Department of Urology Research, Rome, Georgia
  - North Fulton Urology, Roswell, Georgia
  - St. Joseph's, Candler Health System, Savannah, Georgia
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Prairie Medical Associates, Chicago, Illinois
  - Medical and Surgical Specialists, Galesburg, Illinois
  - Special Care Research, Peoria, Illinois
  - Urology of Indiana, LLC, Greenwood, Indiana
  - MMPC Urology, Greenwood, Indiana
  - Metropolitan Urology, Jeffersonville, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - LSUHSC/Stanley Scott Cancer Center, New Orleans, Louisiana
  - Regional Urology LLC, Shreveport, Louisiana
  - Anne Arundel Urology P.A., Annapolis, Maryland
  - Maryland Prostate Center: University of Maryland Medical Center, Baltimore, Maryland
  - Urology Center, PA, Hagerstown, Maryland
  - Mid Atlantic Clinical Research, Rockville, Maryland
  - The Fallon Clinic, Worcester, Massachusetts
  - Wayne Glazier, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Beaumont Medical, Royal Oak, Michigan
  - Mayo Clinic Urology Department, Rochester, Minnesota
  - Park Nicollet Urology, Saint Louis Park, Minnesota
  - Kansas City Urology, PC, Kansas City, Missouri
  - PPS Clinical Research, St Louis, Missouri
  - Urologic Research Center, St Louis, Missouri
  - Sheldon Freeman, Las Vegas, Nevada
  - Urologic Surgeons, Ltd., Reno, Nevada
  - Coastal Urology Associates, Brick, New Jersey
  - Hamilton Urology PA, Hamilton, New Jersey
  - Lawrenceville Urology Associates, Lawrenceville, New Jersey
  - Assoc. Urologic Specialists, Marlton, New Jersey
  - Urology Healthcare Associates, Willingboro, New Jersey
  - Urology Group of New Mexico, Albuquerque, New Mexico
  - Urology Inst. Of New York, Albany, New York
  - William Oberheim, Albany, New York
  - Metropolitan Urologic Services, PC, Elmont, New York
  - Urological Surgeons of Long Island, Garden City, New York
  - University Urology Associates, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - CNY Urology, Oneida, New York
  - Staten Island Urological Research , PC, Staten Island, New York
  - Associated Urologists of CNY, Syracuse, New York
  - Center for Urologic Research WNY, LLC, Williamsville, New York
  - Asheboro Urology, Asheboro, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - The Urology Center, Greensboro, North Carolina
  - Wake Urology, Raleigh, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Odyssey Research, Bismarck, North Dakota
  - Summa Health Care, Akron, Ohio
  - The Urology Group, Cincinnati, Ohio
  - Cleveland Clinic Lerner College of Medicine, Cleveland, Ohio
  - Colombus Urology Research, Columbus, Ohio
  - Urology of Northern Ohio, Elyria, Ohio
  - Southwest Urology, Parma, Ohio
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Urologic Specialists of Oklahoma, Inc., Tulsa, Oklahoma
  - The Corvallis Clinic, Corvallis, Oregon
  - Oregon Urology Specialists, Springfield, Oregon
  - Urologic Associates of Allentown, Allentown, Pennsylvania
  - Urologic Surgery, Bala-Cynwyd, Pennsylvania
  - Urological Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - The Urology Institute, Monroeville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Ginsberg and Harkaway Urology, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - State College Urologic Association, State College, Pennsylvania
  - University Urological Research Institute, Providence, Rhode Island
  - Radiant Research, Greer, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Volunteer Research Group, Knoxville, Tennessee
  - Southeast Urology Network, Memphis, Tennessee
  - Ace Research Specialists, Nashville, Tennessee
  - Center for Urological Treatment, Nashville, Tennessee
  - Urology Associates, Nashville, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Professional Quality Research, Austin, Texas
  - Breco Research, Houston, Texas
  - Urology Consultants, PA, San Antonio, Texas
  - Urology San Antonio Research, PA, San Antonio, Texas
  - Scott and White Clinical Hospital, Temple, Texas
  - Salt Lake City Research, Salt Lake City, Utah
  - Adult and Pediatric Urologists of Northern VA, Alexandria, Virginia
  - Devine Tidewater Urology, Norfolk, Virginia
  - Med Atlantic, Inc (Virginia Urology), Richmond, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Seattle VAMC, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - University of Wisconsin Medical School: Clinical Trials, Madison, Wisconsin
  - St. Michael's Hospital, Milwaukee, Wisconsin
  - Froedtert Memorial Lutheran Hospital Department of Urology, Milwaukee, Wisconsin
  - Wyoming Research Foundation, Cheyenne, Wyoming
- Mexico (19):
  - American British Cowdray Hospital, Mexico City, D. F
  - Centro Medico Dalinde, Mexico City, D. F
  - Hospital General de Mexico, Mexico City, D. F
  - Hospital Regional "Gabriel Mancera", IMSS, Mexico City, D.f,
  - Centro Medico Naval, Mexico City, D.f.
  - Hospital General de Zona No. 1-A, Mexico City, D.f.
  - Clinica Londres, Mexico City, D.f.
  - Hospital Central Militar, SDN, Mexico City, D.f.
  - Hospital Medica Sur, Mexico City, D.f.
  - Hospital de Oncologia CMN Siglo XXI, IMSS, Mexico City, D.f.
  - Hospital General de Zona No. 26, Mexico D.F., Mexico City, D.f.
  - Hospital General Region 1 de Octubre, ISSSTE, Mexico City, D.F
  - Hospital Civil Viejo "Fray Antonio Alcalde", Guadalajara, Jalisco
  - Centro Medico de Occidente-IMSS, Guadalajara, Jalisco
  - Hospital Regional Dr Valentin Gomez Farias, ISSSTE, Guadalajara, Jalisco
  - Hospital Regional de Especialidades, Monterrey, N.l.
  - Hospital Universitario, Monterrey, N.l.
  - Hospital Ignacio Morones Prieto, San Luis Potosí City, S.l.p.
  - Hospital General de Zona con UMF No. 2 San Luis Potosi, San Luis Potosí City, S.l.p.

REFERENCES:
- [Derived] Smith MR, Morton RA, Barnette KG, Sieber PR, Malkowicz SB, Rodriguez D, Hancock ML, Steiner MS. Toremifene to reduce fracture risk in men receiving androgen deprivation therapy for prostate cancer. J Urol. 2013 Jan;189(1 Suppl):S45-50. doi: 10.1016/j.juro.2012.11.016. PMID 23234631
- [Derived] Morgans AK, Hancock ML, Barnette KG, Steiner MS, Morton RA, Smith MR. Racial differences in bone mineral density and fractures in men receiving androgen deprivation therapy for prostate cancer. J Urol. 2012 Mar;187(3):889-93. doi: 10.1016/j.juro.2011.10.136. Epub 2012 Jan 15. PMID 22245322